CLINICAL TRIAL: NCT02631863
Title: A Pilot Study of Photodynamic Therapy (PDT) Using Aminolaevulinic Acid (ALA) in Patients With HPV+ Low Grade Cervical Intraepithelial Neoplasia (LSIL;CIN1)
Brief Title: Aminolaevulinic Acid Photodynamic Therapy for HPV+ Low Grade Cervical Intraepithelial Neoplasia (LSIL;CIN1)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Fudan-Zhangjiang Bio-Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FDZJALA-201510
Record Dates: First submitted 2015-12-12; First posted 2015-12-16 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Cervical Intraepithelial Neoplasia; Low-Grade Squamous Intraepithelial Lesions; Papillomavirus Infections
MeSH Terms: conditions — Uterine Cervical Dysplasia; Squamous Intraepithelial Lesions; Papillomavirus Infections | interventions — 5-aminolaevulinic acid-n-pentylester

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALA (Experimental): Patients will receive 3 topical treatments of aminolaevulinic acid 500mg
  Interventions: Drug: Aminolaevulinic acid
- Placebo (Placebo Comparator): Patients will receive 3 topical treatments of placebo 500mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aminolaevulinic acid — Aminolaevulinic acid with illumination
  Arms: ALA
Drug: Placebo — Placebo with illumination
  Arms: Placebo

SUMMARY:
This trial will study the effectiveness of photodynamic therapy with aminolaevulinic acid for the treatment of patients with HPV+ low grade cervical intraepithelial neoplasia (LSIL;CIN1).

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women, 25-50 years of age
* Diagnosed with LSIL/CIN1 by local pathology (biopsy) and high-risk HPV positive by HC2 assay within the last 3 months
* Satisfactory colposcopy examination (visibility of entire transformation zone and entire lesion margin )
* Meet the following conditions: pregnancy test negative; no pregnancy plan during the trial; no sexuality or reliable contraceptive measures taken since last menstruation to the onset of the study, agreeing to adopt reliable contraceptive measures during the study
* Written informed consent signed

Exclusion Criteria:

* ASC-H (atypical squamous cells, cannot exclude HSIL) or HSIL (high-grade squamous intraepithelial lesions) or AGC (atypical glandular cells) or AIS (adenocarcinoma in situ) on cytology, or malignant cells on cytology or histology, or other suspicion of either micro-invasive or invasive disease
* Invasive carcinoma possibility or lesions extending to the vaginal vault or suspicion of endocervical disease on colposcopy
* Severe pelvic inflammatory disease, severe cervicitis, or other severe gynaecological infection as per clinical examination
* Undiagnosed vaginal bleeding
* With allergic disease at present; known or suspected porphyria; known allergy to ALA or analogues
* With serious cardiovascular, neurologic, psychiatric, endocrine, hematological disease; immunocompromised conditions; patients with malignant tumors
* Hepatic or renal functions abnormal (alanine aminotransferase or aspartate transaminase or total bilirubin > 1.5 upper limit of normal [ULN], or serum creatinine or blood urea nitrogen > 1.5 ULN)
* Pregnancy or nursing
* Previous physical therapy of LSIL/CIN1 after pathologic diagnosis
* Participation in any clinical studies within the last 30 days
* Subjects that the investigators judged to be not suitable to participate the study besides above

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-03-22 (Actual); Primary Completion 2018-11-24 (Actual); Study Completion 2018-11-24 (Actual)

PRIMARY OUTCOMES:
Response rate | 3 months after treatments
  Based on histology, cytology and HPV status. "Response" is defined as: 1) pathology and cytology were both normal; 2) pathology and/or cytology showed low grade and the baseline HPV infection was cleared.
Complete response rate | 3 months after treatments
  Based on histology, cytology and HPV status. "Complete response" is defined as normal pathology, normal cytology and negative HPV.
Clearance of high risk HPV | 3 months after treatments
  Proportion of patients with high risk HPV clearance

CONTACTS AND LOCATIONS:
Overall Officials: Beihua Kong, MD, Principal Investigator — Qilu Hospital of Shandong University; Youzhong Zhang, MD, Principal Investigator — Qilu Hospital of Shandong University; Jining Tao, Study Director — Shanghai Fudan-Zhangjiang Bio-Pharmaceutical Co., Ltd.
Locations (4):
- China (4):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The Obstetrics & Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Women's Hospital School of Medicine Zhejiang University, Hangzhou, Zhejiang